CLINICAL TRIAL: NCT00717704
Title: A Phase I Study of Ixabepilone Combined With Dasatinib in Patients With Solid Tumors
Brief Title: Solid Tumors Using Ixabepilone and Dasatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WCI-2007-528
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2012-05

CONDITIONS: Solid Tumor
Keywords: Malignant solid tumor; Phase 1; Dose escalation; Metastatic or locally advanced/unresectable; Disease progression through standard therapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ixabepilone; Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All participants will receive ixabepilone by vein once every three weeks as well as dasatinib by mouth once daily. All participants will receive the study drugs at a baseline dose. If the side effects are minimal and tolerable, the next cycle of study drugs will be given at same dosage. If side effects are intolerable, then the dose will be lowered.
  Interventions: Drug: ixabepilone; Drug: Dasatinib

INTERVENTIONS:
Drug: ixabepilone — by vein once every 3 weeks
  Other Names: ixempra
Drug: Dasatinib — by mouth once daily
  Other Names: Sprycel; BMS-354825

SUMMARY:
Patients are being asked to take part in this study because they have been diagnosed with an advanced solid tumor that is not responding to standard treatments. This study will find the highest dose of ixabepilone and dasatinib in combination that can be given without causing severe side effects.

Both ixabepilone and dasatinib have individually been tested in many (several thousand) patients, however the combination of the two drugs has not yet been tested in humans.

All patients who will take part in this study will receive combined drug therapy of dasatinib and ixabepilone. Dasatinib is a pill that is taken by mouth. Ixabepilone is a medicine that will be given by vein (IV).

All participants will receive ixabepilone by vein once every three weeks as well as dasatinib by mouth once daily.

ELIGIBILITY:
Inclusion Criteria:

* Have a solid tumor malignancy that is metastatic or locally advanced/unresectable
* Progression through standard therapy
* Histological documentation of cancer
* Must be off prior chemotherapy or radiation therapy for at least 3 weeks
* Must have adequate organ and marrow function prior to the start of study treatment as defined by the protocol
* Must be able to swallow oral medication (dasatinib must be swallowed whole)
* Must be available for protocol-required follow-up

Exclusion Criteria:

* Patients with a malignancy (other than the one treated in this study) which required radiotherapy or systemic therapy within the past 5 years
* Symptomatic brain metastasis that is either untreated or uncontrolled by surgery and or radiotherapy
* A known, prior, severe (NCI CTC Grade 3/Grade 4) history of hypersensitivity reaction to a drug formulated in Cremophor (polyoxyethylated castor oil)
* A serious, uncontrolled medical disorder or active infection including pericardial or pleural effusion of any grade,uncontrolled or significant cardiovascular disease,a bleeding disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The primary outcome is to determine the safety and toxicity of ixabepilone and dasatinib in combination in patients with metastatic or locally advanced/unresectable solid tumors that have progressed through standard therapy. | From study start until completion of study followup. This can vary greatly between patients, but on average patients received treatment for 4 cycles (12 weeks).
  While on the drug combination, patients will be seen in the clinic every 3 weeks. These visits will assess the safety and tolerablility of the drug regimen. The drug combination continues until disease progression or unacceptable toxicity. When one of those two events occurs, the patient enters the followup phase. During the followup phase, the patient will return to the clinic every 4 weeks until drug-related toxicities resolve.

SECONDARY OUTCOMES:
The secondary outcome is to evaluate tumor response as a preliminary assessment of clinical activity. | From start of the study until completion of the drug regimen. This can vary greatly between patients, but on average patients received treatment for 4 cycles (12 weeks).
  Disease status will be monitored via diagnostic imaging every other cycle (every six weeks) until the patient is finished with drug combination. The drug combination continues until disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Swain, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Cancer Institute, Washington D.C., District of Columbia, United States